CLINICAL TRIAL: NCT03698955
Title: A Randomized, Cross-Over Trial on the Effects of a Low-Fat Vegan Diet Versus a Mediterranean Diet on Body Weight
Brief Title: Low-Fat Vegan Diet Versus a Mediterranean Diet on Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00029777
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-02

CONDITIONS: Overweight; Obesity; Insulin Resistance
Keywords: Plant-based diet; Mediterranean diet; Vegan diet; Metabolism; Insulin sensitivity; Cholesterol; Advanced glycation end-products
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance | interventions — Diet, Plant-Based; Diet, Vegan; Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plant-based diet (Active Comparator): The diet group will be asked to follow a low-fat, vegan diet for 16 weeks.
  Interventions: Other: Plant-based diet
- Mediterranean diet (Active Comparator): The diet group will be asked to follow a Mediterranean diet for 16 weeks.
  Interventions: Other: Mediterranean Diet

INTERVENTIONS:
Other: Plant-based diet — Weekly instructions will be given to the participants in the intervention group about following the vegan diet.
  Other Names: Vegan diet
  Arms: Plant-based diet
Other: Mediterranean Diet — Weekly instructions will be given to the participants in the intervention group about following the Mediterranean diet.
  Arms: Mediterranean diet

SUMMARY:
This randomized, cross-over trial aims to assess changes in body weight, plasma lipids, insulin sensitivity, and postprandial metabolism with a low-fat, plant-based diet and a Mediterranean diet, both followed for 4 months.

DETAILED DESCRIPTION:
In a 36-week cross-over trial, overweight adults will consume a low-fat vegan diet and a Mediterranean diet in two separate 16-week phases. Changes in body weight will be the primary dependent variable. In addition, plasma lipid concentrations, insulin sensitivity, and postprandial metabolism will also be assessed and changes over time will be compared between the two diets.

Participants will be randomly assigned to start either a low-fat vegan diet or a Mediterranean diet for 16 weeks. Both groups will receive weekly classes and support, and will be asked to make no changes to their exercise patterns for the study period. After a 4-week washout period, participants will cross over to the second dietary intervention for another 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age ≥18 years of age
* Body mass index 28-40 kg/m2

Exclusion Criteria:

* Diabetes mellitus type 1, history of any endocrine condition that would affect body weight, such as thyroid disease, pituitary abnormality, or Cushing's syndrome
* Smoking during the past six months
* Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
* Use of recreational drugs in the past 6 months
* Use within the preceding six months of medications that affect appetite or body weight, such as estrogens or other hormones, thyroid medications (unstable dose within the preceding 6 months), systemic steroids, antidepressants (tricyclics, MAOIs, SSRIs), antipsychotics, lithium, anticonvulsants, appetite suppressants or other weight-loss drugs, herbs for weight loss or mood, St. John's wort, ephedra, beta blockers
* Pregnancy or intention to become pregnant during the study period, as verified by self--- - Unstable medical or psychiatric illness
* Evidence of an eating disorder
* Likely to be disruptive in group sessions
* Already following a low-fat vegan diet or Mediterranean diet
* Lack of English fluency
* Inability to maintain current medication regimen
* Inability or unwillingness to participate in all components of the study
* Intention to follow another weight-loss method during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Body weight | Change in body weight from Baseline at 4 months
  Body weight will be assessed at the baseline and at the completion of both interventions.
Plasma lipids | Change in plasma cholesterol, triglycerides, and HbA1c from Baseline at 4 months
  Plasma cholesterol, triglycerides, and HbA1c will be measured in a fasting state.
Insulin sensitivity | Change in insulin sensitivity from Baseline at 4 months
  Insulin sensitivity will be assessed by the HOMA index.
Metabolism | Changes in metabolism from Baseline at 4 months
  Participants will be asked to report to the laboratory within 60 minutes of waking and after a 12-hour fast. Following 30 minutes of quiet rest in a dimly lit room, pulse, respiratory rate, and body temperature will be measured. REE will be measured for 20 minutes through indirect calorimetry (Cosmed Quark RMR, Chicago, IL) utilizing a ventilated hood system. The laboratory temperature will be maintained at 23 degrees C throughout, and precautions will be taken to minimize any disturbances that could affect the metabolic rate.
  For premenopausal women, measures will be timed so as to occur in the luteal phase of the menstrual cycle. Postprandial metabolism will be measured for three hours after the standard meal.

SECONDARY OUTCOMES:
Levels of Advanced Glycosylation Endproducts (AGEs) | Change in Advanced Glycosylation Endproducts (AGEs) from Baseline at 4 months
  An AGE reader will be used to measure the Levels of the AGEs in the skin
Endothelial function | Change in Endothelial function from Baseline at 4 months
  Endothelial function will be measured using the EndoPAT.
Microbiome analysis | Change in Microbiome from Baseline at 4 months
  Microbiome analysis will be performed from participant-provided stool sample. Anticipated changes in the dietary intervention group include changes in the microbiome composition that correlate with changes in insulin sensitivity.
Dietary Advanced Glycation End Products (AGEs) | 16 weeks
  Explore the effectiveness of a vegan diet in reducing dietary AGEs.
PDI, hPDI, uPDI | 16 weeks
  Assess the total plant-based index (PDI), healthy PDI, and unhealthy PDI, and their relationship with weight loss.
Ultraprocessed foods | 16 weeks
  The consumption of ultraprocessed foods will be assessed, using the NOVA classification, at baseline and 16 weeks.
Carbon Footprint | 16 weeks
  The greenhouse gas emissions (GHGE) and cumulative energy demand (CED) will be assessed, using the database of Food Impacts on the Environment for Linking to Diets (dataFIELD) and What We Eat In America (WWEIA) database, at baseline and 16 weeks.
Food costs | 16 weeks
  Food costs will be assessed, using the U.S. Department of Agriculture Thrifty Food Plan, 2021, at baseline and 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Neal Barnard, Principal Investigator — Physicians Committee for Responsible Medicine
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kahleova H, Smith R, Fischer I, Brennan H, Znayenko-Miller T, Holubkov R, Barnard ND. Plant-based dietary index on the Mediterranean and a vegan diet: a secondary analysis of a randomized, cross-over trial. Front Nutr. 2025 Nov 19;12:1666807. doi: 10.3389/fnut.2025.1666807. eCollection 2025. PMID 41346691
- [Derived] Kahleova H, Maracine C, Himmelfarb J, Jayaraman A, Znayenko-Miller T, Holubkov R, Barnard ND. Dietary acid load on the Mediterranean and a vegan diet: a secondary analysis of a randomized, cross-over trial. Front Nutr. 2025 Jun 25;12:1634215. doi: 10.3389/fnut.2025.1634215. eCollection 2025. PMID 40635898
- [Derived] Kahleova H, Znayenko-Miller T, Motoa G, Eng E, Prevost A, Uribarri J, Holubkov R, Barnard ND. Dietary advanced glycation end-products and their associations with body weight on a Mediterranean diet and low-fat vegan diet: a randomized, cross-over trial. Front Nutr. 2024 Aug 8;11:1426642. doi: 10.3389/fnut.2024.1426642. eCollection 2024. PMID 39176029
- [Derived] Kahleova H, McCann J, Alwarith J, Rembert E, Tura A, Holubkov R, Barnard ND. A plant-based diet in overweight adults in a 16-week randomized clinical trial: The role of dietary acid load. Clin Nutr ESPEN. 2021 Aug;44:150-158. doi: 10.1016/j.clnesp.2021.05.015. Epub 2021 May 29. PMID 34330460
- [Derived] Barnard ND, Alwarith J, Rembert E, Brandon L, Nguyen M, Goergen A, Horne T, do Nascimento GF, Lakkadi K, Tura A, Holubkov R, Kahleova H. A Mediterranean Diet and Low-Fat Vegan Diet to Improve Body Weight and Cardiometabolic Risk Factors: A Randomized, Cross-over Trial. J Am Nutr Assoc. 2022 Feb;41(2):127-139. doi: 10.1080/07315724.2020.1869625. Epub 2021 Feb 5. PMID 33544066